CLINICAL TRIAL: NCT06272565
Title: An Approach of Exploring the Mechanism of the Interaction Between Metabolic Disorders and NLPR3 Inflammasome Activation in DR Inflammatory Damage Based on Metabolomics Methods
Brief Title: Exploring the Interaction Between Metabolic Disorders and NLPR3 Inflammasome Activation in DR Inflammatory Damage
Acronym: DR
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023KYPJ292
Record Dates: First submitted 2024-02-01; First posted 2024-02-22 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; Anti-vascular Endothelial Growth Factor
Keywords: Diabetic retinopathy; metabolomics; NLPR3; Diabetic Macular edema; Anti-vascular endothelial growth factor
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and aqueous humor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CON(Non diabetes control group): Non diabetes patients undergoing phacoemulsification surgery
- NDR(Non diabetes retinopathy diabetes patients): Non DR diabetes patients undergoing phacoemulsification surgery
- NPDR (non proliferative diabetes retinopathy): DR patients with no sign of any neovascularization suggested by fluorescein sodium angiography and receiving intravitreal injection surgery
- PDR (proliferative diabetes retinopathy): DR patients with neovascularization suggested by fluorescein sodium angiography and receiving intravitreal injection surgery

SUMMARY:
Diabetic retinopathy (DR) is one of the most serious microvascular complications of diabetes. Early diagnosis and treatment of diabetes is the key to prevent visual impairment in DR patients. This study aims to use a non-targeted metabolomics detection technique combined with ultra-high performance liquid chromatography time-of-flight mass spectrometry to analyze the metabolomics profile in aqueous humor sample of DR patents, and further explore the mechanism of the relationship between differential metabolites and their metabolic pathways with NLRP3 activation in DR inflammatory damage. DR patients with macular edema will receive anti-vascular endothelial growth factor (anti-VEGF) treatment; these patients will be divided into two groups: responders group and non-responders group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 40 years old.
2. CON (non diabetes control group)：patients undergoing phacoemulsification surgery.
3. NDR (non diabetes retinopathy diabetes patients): patients with diabetes history and undergoing phacoemulsification surgery.
4. NPDR (non proliferative diabetes retinopathy): patients with history of diabetes, fundus microangiopathy shown by fundus fluorescein angiography, including microangioma, hard exudation, wadding exudation and other non proliferative diabetes retinopathy signs, and did not receive invasive ophthalmic treatment within 3 months.
5. PDR (proliferative diabetes retinopathy): patients with a history of diabetes, fundus neovascular lesions shown by fundus fluorescein angiography, and did not receive invasive ophthalmic treatment within 3 months.
6. Patients voluntarily signed informed consent.

Exclusion Criteria:

1. CON (non diabetes control group)：patients with a history of other ophthalmic operations.
2. NDR (non diabetes retinopathy diabetes patients): patients with fundus changes of diabetes retinopathy or other ophthalmic surgery history.
3. NPDR (non proliferative diabetes retinopathy): patients with fundus neovascular lesions shown by fundus fluorescein angiography.
4. PDR (proliferative diabetes retinopathy):patients undergoing vitrectomy。
5. Patients with active ocular inflammation, high myopia, pregnancy.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. CON (non diabetes control group)：Non diabetes patients undergoing phacoemulsification surgery.
  2. NDR (non diabetes retinopathy diabetes patients): Non DR diabetes patients undergoing phacoemulsification surgery.
  3. NPDR (non proliferative diabetes retinopathy): DR patients with no sign of any neovascularization suggested by fluorescein sodium angiography and receiving intravitreal injection surgery.
  4. PDR (proliferative diabetes retinopathy): DR patients with neovascularization suggested by fluorescein sodium angiography and receiving intravitreal injection surgery.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-07-03 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Untargeted metabolomics for metabolic profile using UHPLC/MS | 24 weeks
  Aqueous humor samples in DR patients will be analysed to putatively identify metabolic profile by comparison with control samples using ultra-high performance liquid chromatography-high resolution mass spectrometer (UHPLC/MS). UHPLC/MS analysis allows the simultaneous high-resolution measurement of a broad range of metabolites, hence the untargeted nature of the analysis.
  For the UHPLC/MS results, perform normalization, standardization, and log transformation, then compare the metabolite differences between groups.
  Multivariate statistical analysis and Partial least squares discriminant analysis included in the mass spectrometry software will be used to analyse UHPLC/MS results to identify metabolites that best discriminate between DR and control conditions. The evaluation of significant metabolite results is based on: P-value and Fold change.

SECONDARY OUTCOMES:
Best-corrected visual acuity | 24 weeks
  Best-corrected visual acuity at baseline and 24 weeks follow-up
Central subfield thickness | 24 weeks
  Central subfield thickness at baseline and 24 weeks follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No